CLINICAL TRIAL: NCT05062096
Title: Characterization of NK Cells Under First Line Advanced Therapy Either as Curative Therapy for Metastatic Melanoma or as Adjuvant Therapy for High-risk of Recurrence
Acronym: NAKIMEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Société de Dermatologie Française (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP200196
Record Dates: First submitted 2021-05-17; First posted 2021-09-30 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Melanoma
Keywords: melanoma; NK cells; targeted therapies; immunotherapies
MeSH Terms: conditions — Melanoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: BRAF-mutated metastatic patients treated with 1st line targeted therapy (Other): BRAF-mutated metastatic patients treated with 1st line targeted therapy
  Interventions: Other: Blood samples; Other: Skin biopsy
- Group 2: Metastatic patients treated with 1st line immunotherapy (Other): Metastatic patients treated with 1st line immunotherapy
  Interventions: Other: Blood samples; Other: Skin biopsy
- Group 3: BRAF-mutated patients treated with adjuvant targeted therapy (Other): BRAF-mutated patients treated with adjuvant targeted therapy
  Interventions: Other: Blood samples; Other: Skin biopsy
- Group 4: Patients treated with adjuvant immunotherapy (Other): Patients treated with adjuvant immunotherapy
  Interventions: Other: Blood samples; Other: Skin biopsy

INTERVENTIONS:
Other: Blood samples — Blood samples at each protocol visit, T and NK cell analysis
Other: Skin biopsy — Biopsy of the skin lesion (optional)

SUMMARY:
Cutaneous melanoma is a tumor with a serious evolution if its initial diagnosis is late. Since 2011, the treatment of advanced forms involves two therapeutic approaches : targeted therapies (BRAF and MEK inhibitors) if the tumor carries a BRAF mutation or immunotherapies (anti-PD1, anti-CTLA-4) regardless of tumor BRAF mutation status. Current data support the hypothesis that combinations of agents targeting the tumor and its environment will be required for durable responses in the majority of patients. Investigators will study the role of NK lymphocytes in tumor immunosurveillance in patients undergoing first-line innovative therapy with metastatic melanoma or at high-risk of recurrence.

DETAILED DESCRIPTION:
Natural Killer (NK) lymphocytes are cytotoxic effectors of the innate immune response that are involved in different phases of tumor immunosurveillance. These lymphocytes are activated upon contact with tumor cells and exert direct cytotoxic activity without prior immunization. Activated NK lymphocytes produce cytokines, including IFN-γ and TNF-α, which induce and maintain an activation of the adaptive immune response by CD8+ lymphocytes. Numerous studies in various experimental tumor models highlight the role of NK cells in the control of metastasis.

Our previous work has shown that NK cells infiltrate primary melanomas, that metastatic patients have altered blood NKs, and furthermore, that chemotherapy modulates their functional status. Investigators also observed a particular distribution of gene polymorphisms encoding NK activating receptors of stage IV melanoma patients compared to healthy donors. Finally, the investigator described a novel population of NK lymphocytes in metastatic lymph nodes draining melanoma NK cell activation is regulated by a balance between activating receptors (NKG2D, NCR) and inhibitory receptors that bind to modulatory classical and non-classical HLA-I molecules (HLA-E and G). More recently it has been shown that Lc NKs also express checkpoint receptors including CD96/TIGIT, NKG2A, TIM3 and PD-1 (the latter 2 are present on LcTs) that negatively modulate NK activation. The possibility of activating the lytic and secretory function of Lc NKs by interfering with these receptors may represent an alternative yet to be explored in immunotherapy treatments.

More recently, th investigator have developed a program to understand the interactions between tumor mutational profile, treatment with targeted therapies and NK immunogenicity. the investigator have a panel of melanoma lines with and without the BRAF V600E mutation and vemurafenib resistant variants have been obtained from some mutated lines. the investigator evaluated the impact of treatment and resistance to BRAF inhibition on Lc NK recognition and lysis. yhe investigator showed that a BRAF inhibitor, vemurafenib, decreased membrane and soluble expression of MICA/B and ULBP2, ligands for NKG2D, an activating receptor present on Lc NKs and certain populations of Lc T cells, in all BRAF mutated lines treated. For 6 of the 7 mutated lines, modulations of NK ligands expression by vemurafenib correlated with a slight decrease in NK cytotoxic functions.

Vemurafenib-resistant (R) variants were generated and their characteristics were compared to those of sensitive (S) lines. The acquisition of resistance to vemurafenib induces a significant increase in NK functions (IFNg secretion and target lysis). The responsible mechanisms involve both the expression of NK receptor ligands and the modulation of death domain receptors (Fas, TRAILRII). Transcriptome analyses reveal different targets of interest in the three pairs of S/R melanoma lines carrying the BRAF V600E mutation and distinct additional mutations (submitted manuscript).

Based on our recent results our hypothesize that Lc NKs are important players in tumor immunosurveillance during current treatments of melanoma patients. Immunotherapy approaches targeting these effectors may be of interest in combinations with targeted therapies or immunotherapies. The frequency of intratumoral Lc NKs has been shown to correlate with the presence of stimulatory dendritic cells and this environment is required for a response to anti-PD1 immunotherapy. Innovative antibodies are being developed to activate the antitumor functions of NK cells

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years
* Histologically confirmed melanoma patient
* Patient for whom treatment by targeted therapy or immunotherapy is prescribed as an adjuvant or curative treatment
* In the case of adjuvant treatment, the tumor must be completely removed
* Patient included in the Ric-Mel cohort
* Patient informed of the objectives and modalities of the study and having received the information form and having given his/her written consent to participate in the research
* Patient affiliated to a social security system

Exclusion Criteria:

* Patient already treated medically for melanoma
* Palliative care patient management
* Pregnant or breastfeeding women
* Patient under guardianship or curatorship
* refusal of the patient to participate in the study, or refusal of the patient to allow a portion of his/her previously collected skin sample to be used in the present research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-02 (Estimated)

PRIMARY OUTCOMES:
characterize lymphoid cells, in particular NK lymphocytes, LcTs before and during a first line of curative or adjuvant treatment by targeted therapy or immunotherapy in order to identify early markers of response/resistance to treatment. | Before the start of treatment and after 3-4 weeks
  NK cells are recovered from blood samples taken before the start of treatment and after 3-4 weeks

SECONDARY OUTCOMES:
Characterize lymphoid cells before and during a first line of curative or adjuvant treatment with targeted therapy or immunotherapy to identify late markers of response/resistance to treatment. | From Mont 2-Month 3 to Mmonth 6
  NK cells are recovered from blood samples taken at 2-3 months to 6 of treatment Late changes from Month2-Month 3 to Month 6 in the expression of membrane or soluble markers of NK or LcT cells during treatment and according to treatment groups (targeted therapy or immunotherapy used in a curative or an adjuvant setting).
Evaluate the association between soluble or membrane markers modified during treatment and clinical evolution | During treatment up to 6 month
  analysis of soluble or membrane markers altered during treatment as a function of responders and non-responders according to RECIST 1.1 criteria.
Immunohistochemical analysis of markers of interest on primary tumors and/or metastases at baseline and during treatment if possible and according to the response to treatment | Before the start of treatment and during treatment up to 6 month
  Tumor biopsy analysis to Identification of tumor markers or combination of tumor markers whose expression is associated with response or resistance to therapy according to RECIST 1.1. If sequential biopsies are obtained in patients with skin metastases, investigation of an association between tumor phenotype in the microenvironment at S3-S4 of treatment and response to treatment
Assess the predictive capacity of soluble tumor markers in blood cells before the beginning of the treatment on the clinical evolution | Before the start of treatment
  Blood analysis evaluat soluble and membrane markers at baseline and during treatment as a function of treatment response
Comparison of soluble or membrane markers modified according to the treatment | During treatment up to 6 months
  Cellular analysis to see modification of the expression of membrane markers (+/- 30% of expression of the marker or Mean Fluorescence) or soluble markers (+/- 20% of expression of the marker) of NK or LcT cells during the treatment and according to the treatment received: targeted therapy or immunotherapy
Comparison of soluble or membrane markers modified according to the presence or not of metastasis | During treatment up to 3 months
  Cellular analysis to study modification of the expression of membrane markers (+/- 30% of expression of the marker or of the Mean Fluorescence) or soluble markers (+/- 20% of expression of the marker) of NK or LcT cells during the treatment and according to the presence or not of metastasis at the inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Eve Maubec, PhD, Principal Investigator — Assistance Public Hôpitaux de Paris

REFERENCES:
- [Background] Frazao A, Colombo M, Fourmentraux-Neves E, Messaoudene M, Rusakiewicz S, Zitvogel L, Vivier E, Vely F, Faure F, Dreno B, Benlalam H, Bouquet F, Savina A, Pasmant E, Toubert A, Avril MF, Caignard A. Shifting the Balance of Activating and Inhibitory Natural Killer Receptor Ligands on BRAFV600E Melanoma Lines with Vemurafenib. Cancer Immunol Res. 2017 Jul;5(7):582-593. doi: 10.1158/2326-6066.CIR-16-0380. Epub 2017 Jun 2. PMID 28576831
- [Background] Martinez EA, Shore A, Colantuoni E, Herzer K, Thompson DA, Gurses AP, Marsteller JA, Bauer L, Goeschel CA, Cleary K, Pronovost PJ, Pham JC. Cardiac surgery errors: results from the UK National Reporting and Learning System. Int J Qual Health Care. 2011 Apr;23(2):151-8. doi: 10.1093/intqhc/mzq084. Epub 2011 Jan 10. PMID 21224272
- [Background] Messaoudene M, Fregni G, Enot D, Jacquelot N, Neves E, Germaud N, Garchon HJ, Boukouaci W, Tamouza R, Chanal J, Avril MF, Toubert A, Zitvogel L, Rusakiewicz S, Caignard A. NKp30 isoforms and NKp46 transcripts in metastatic melanoma patients: Unique NKp30 pattern in rare melanoma patients with favorable evolution. Oncoimmunology. 2016 Mar 10;5(12):e1154251. doi: 10.1080/2162402X.2016.1154251. eCollection 2016. PMID 28123867
- [Background] Messaoudene M, Fregni G, Fourmentraux-Neves E, Chanal J, Maubec E, Mazouz-Dorval S, Couturaud B, Girod A, Sastre-Garau X, Albert S, Guedon C, Deschamps L, Mitilian D, Cremer I, Jacquelot N, Rusakiewicz S, Zitvogel L, Avril MF, Caignard A. Mature cytotoxic CD56(bright)/CD16(+) natural killer cells can infiltrate lymph nodes adjacent to metastatic melanoma. Cancer Res. 2014 Jan 1;74(1):81-92. doi: 10.1158/0008-5472.CAN-13-1303. Epub 2013 Nov 13. PMID 24225017
- [Background] Sastre J, Diaz-Beveridge R, Garcia-Foncillas J, Guardeno R, Lopez C, Pazo R, Rodriguez-Salas N, Salgado M, Salud A, Feliu J. Clinical guideline SEOM: hepatocellular carcinoma. Clin Transl Oncol. 2015 Dec;17(12):988-95. doi: 10.1007/s12094-015-1451-3. Epub 2015 Nov 25. PMID 26607931
- See also: Minimally Invasive Treatments for Liver Cancer, Updates in Liver Cancer — https://www.intechopen.com/books/updates-in-liver-cancer/minimally-invasive-treatments-for-liver-cancer